CLINICAL TRIAL: NCT03167086
Title: "Empowered Relief" Single Session Pain Psychology Treatment: Comparative Efficacy & Mechanisms
Brief Title: Single Session Pain Psychology Treatment: Comparative Efficacy & Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Beth Darnall, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT008561 (NIH)
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The design is a randomized 3-arm study comprised of 2 active psychological treatments (ER & CBT) and a health education (HE) arm that controls for time and attention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Principal Investigators and Statisticians performing analyses will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Session Skills-Based Pain Psychology Class (Experimental): "Empowered Relief (ER)": A single-session skills-based approximately 2-hr group intervention for chronic pain.
  Interventions: Behavioral: "Empowered Relief" (ER)
- Cognitive Behavioral Therapy (CBT) (Active Comparator): 8-week Manualized Pain-CBT Group Intervention will be delivered by PhD-level psychotherapists (3 in total).
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Health Education (HE) (Active Comparator): The active control treatment arm consists only of Health Education and has no psychological treatment components. It is a 2-hour HE class matched to the single-session psychological experimental arm (ER) on 4 important factors: duration, structure, format and site.
  Interventions: Behavioral: Health Education (HE)

INTERVENTIONS:
Behavioral: "Empowered Relief" (ER) — "Empowered Relief (ER)": A single-session skills-based approximately 2-hr group intervention to treat chronic pain.
  Format of intervention: Therapist-delivered PowerPoint presentation with experiential exercises. Experienced senior level psychologist and two (2) additional doctoral level psychologists will conduct the ER sessions.
  Content of intervention: ER Participants have the 'ER Relaxation Resource' app (guided relaxation audiofile) loaded on their apple or android electronic device.
  Arms: Single Session Skills-Based Pain Psychology Class
Behavioral: Cognitive Behavioral Therapy (CBT) — Format of intervention: 8-week Manualized Pain-CBT Group Intervention will be delivered by PhD-level psychotherapists (3 in total). The group is run weekly for 8 consecutive classes. Each class is 2 hours with a midpoint break (16 hours total intervention time).
  Content of intervention: The protocol and materials were developed with funding from NIH/NCCAM R01 AT006226 (Dan Cherkin, PI) [1& 2], and include content from a pain-CBT program developed by Drs. Ehde, Dillworth, and Turner [3].
  Participants receive a workbook with homework and a copy of The Pain Survival Guide: How to reclaim your life © 2005 by Turk & Winter [4] for optional reading.
  Arms: Cognitive Behavioral Therapy (CBT)
Behavioral: Health Education (HE) — Format of intervention: The HE class will be instructor taught and will involve a PowerPoint presentation and handouts. Two additional providers will be identified and trained to conduct the sessions. Selected instructors will have substantial health education experience.
  Content of intervention: HE content will include basic information such as nutrition and interacting with the healthcare system; these relatively 'inert' topics are unlikely to impart any specific effects typically found with a true psychobehavioral intervention.
  Arms: Health Education (HE)

SUMMARY:
This study aims to compare the efficacy of a single session psychological treatment, "Empowered Relief" (ER), with the current standard of care, group Cognitive Behavioral Therapy (CBT) specifically on individuals with chronic low back pain who have pain-specific distress as indexed by pain catastrophizing scores.

DETAILED DESCRIPTION:
This is a randomized 3-arm study comprised of 2 active psychological treatments (ER & CBT) and a health education (HE) arm that controls for time and attention. Study goals are to provide scientific evidence to demonstrate the efficacy of ER, and also provide a comparison of said efficacy against the current gold standard group treatment for PC -- manualized 8-session pain-CBT.

ELIGIBILITY:
Inclusion Criteria:

* Axial low back pain without radicular symptoms
* Pain duration ≥ 6 months (per recent NIH Task Force on Research Standards for Chronic Low Back Pain based on participant self-report
* Average pain intensity ≥4/10 for the past month at screening visit
* English fluency
* Males and females 18-70 years of age
* Pain Catastrophizing Score (PCS) ≥20

Exclusion Criteria:

* Gross cognitive impairment
* Active suicidal ideation or severe depression
* Previous attendance in the active treatment groups (any ER classes ever taken or CBT in the past 3 years)
* Participating in any interventional research study or completed participation in the last 2 months; enrollment in an observational study is acceptable
* Current substance abuse
* Clear likelihood to disrupt fellow class participants (e.g., personality disorder) at the discretion of the study team

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Trait Pain Catastrophizing (Trait PC) | 3 months Post-Treatment
  Change in Trait Pain Catastrophizing (Trait PC) from baseline to 3 months post-treatment across all treatment groups

SECONDARY OUTCOMES:
Trait PC at 6 months Post-treatment | 6 months Post-Treatment
  Change in Trait Pain Catastrophizing (Trait PC) from baseline to 6 months post-treatment across all treatment groups
PROMIS Measures at 3 months Post-treatment | 3 months Post-Treatment
  Change in score of PROMIS domains for chronic pain - including pain intensity, physical functioning, and emotional functioning - from baseline to post-treatment 3 months across all three treatment groups
Actigraphy for function and sleep | Several time frames from baseline to 3 months Post-Treatment
  Change in activity & sleep measures from baseline to post-treatment across all treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Beth Darnall, PhD, Principal Investigator — Stanford University; Sean Mackey, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Systems Neuroscience and Pain Lab, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Stoelb, B., Balderson, B., Turner, J.A., Mind-Body Approaches to Pain Management (MAP) Study: CBT Therapist Manual. 2012, Seattle, WA: Group Health Research Institute. (Developed with funding from NIH/NCCAM R01 AT006226; Dan Cherkin, PhD, Principal investigator).
- [Background] 2. Stoelb, B., Balderson, B., Turner, J.A., Mind-Body Approaches to Pain Management (MAP) Study: CBT Patient Workbook. 2012, Seattle, WA: Group Health Research Institute (Developed with funding from NIH/NCCAM R01 AT006226; Dan Cherkin, PhD, Principal Investigator).
- [Background] 3. Ehde, D.M., Dillworth, T. M., & Turner, J.A. , Cognitive-Behavioral Therapy Manual for the Telephone-Delivered Intervention for Pain Study (Unpublished treatment manual). 2012.
- [Background] 4. Turk, D.C., Winter, F., The Pain Survival Guide: How to reclaim your life. 2005, Washington, D.C.: American Psychological Association.
- [Derived] Darnall BD, Roy A, Chen AL, Ziadni MS, Keane RT, You DS, Slater K, Poupore-King H, Mackey I, Kao MC, Cook KF, Lorig K, Zhang D, Hong J, Tian L, Mackey SC. Comparison of a Single-Session Pain Management Skills Intervention With a Single-Session Health Education Intervention and 8 Sessions of Cognitive Behavioral Therapy in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2113401. doi: 10.1001/jamanetworkopen.2021.13401. Erratum In: JAMA Netw Open. 2022 Apr 1;5(4):e229739. doi: 10.1001/jamanetworkopen.2022.9739. PMID 34398206
- [Derived] Darnall BD, Ziadni MS, Roy A, Kao MC, Sturgeon JA, Cook KF, Lorig K, Burns JW, Mackey SC. Comparative Efficacy and Mechanisms of a Single-Session Pain Psychology Class in Chronic Low Back Pain: Study Protocol for a Randomized Controlled Trial. Trials. 2018 Mar 6;19(1):165. doi: 10.1186/s13063-018-2537-3. PMID 29510735